CLINICAL TRIAL: NCT03438032
Title: Identifying Unique Pathogenic Macrophages in Systemic Sclerosis-ILD Using High Throughput Single-cell RNA-Seq
Brief Title: Identifying Unique Pathogenic Macrophages in Systemic Sclerosis-ILD
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Cara J. Gottardi, Associate Professor of Medicine, Northwestern University
Other Study IDs: SP0044402
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Fibrosis Lung; Systemic Sclerosis
MeSH Terms: conditions — Pulmonary Fibrosis; Scleroderma, Systemic | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SSc-ILD: SSc-ILD subjects will be defined by those who fulfill 2013 American College of Rheumatology SSc criteria and have forearm modified Rodnan skin scores (mRSS) ≥1 (a validated, semi-quantitative scoring system for dermal fibrosis) and clinically relevant SSc-interstitial lung disease (ILD). A subject will be defined as having ILD if they have radiographic evidence for ILD and a forced vital capacity <70% on pulmonary function test (PFT).
  Interventions: Diagnostic Test: Bronchoscopy with lavage
- Control: Healthy control subjects recruited from the Northwestern community will complete demographic and basic medical forms to ensure health
  Interventions: Diagnostic Test: Bronchoscopy with lavage

INTERVENTIONS:
Diagnostic Test: Bronchoscopy with lavage — During an elective bronchoscopy procedure, the bronchoscope will be wedged into an affected lung segment guided by CT scanning. When involved an anterior segment will be used to maximize return. After wedging the bronchoscope, 120ml of sterile 0.09% normal saline will be instilled. Up to 40-60 mL of BAL fluid will be obtained for analysis during each sampling.

SUMMARY:
Alveolar macrophages isolated from bronchoalveolar lavage (BAL) fluid from systemic sclerosis (SSc) patients with clinically significant lung fibrosis will be studied at baseline and at 6 months after enrollment to assess longitudinally the presence and persistence of an emergent, pro-fibrotic alveolar macrophage population, using single cell RNA-Seq technology to measure the individual transcriptome from each cell.

DETAILED DESCRIPTION:
Using cutting-edge single cell RNA-Seq technology, we will identify in the BAL fluid of subjects of SSc-ILD emerging pathogenic cell populations in the lung that were previously unrecognized using standard RNA-Seq and microarray technologies, which lack the resolution to analyze transcriptomes of individual cells. Alveolar macrophages isolated from bronchoalveolar lavage (BAL) fluid from SSc patients with clinically significant lung fibrosis will be studied at baseline and at 6 months after enrollment to assess longitudinally the presence and persistence of an emergent, pro-fibrotic alveolar macrophage population.

Subjects with SSc-ILD will be recruited from the Scleroderma Program. We will recruit adults who fulfill 2013 American College of Rheumatology (ACR) SSc criteria and clinically relevant SSc-interstitial lung disease. Patients will undergo bronchoscopy with bronchoalveolar lavage at month 0 and then at month 6. Healthy control subjects will complete demographic and basic medical forms to ensure health. Pertinent clinical data will be downloaded from the Enterprise Data Warehouse, an electronic database in use at Northwestern that was designed to aggregate and store patient data from various medical systems, or through manual chart review, and entered into a RedCap database created specifically for this project.

During an elective bronchoscopy procedure in SSc and healthy control subjects the bronchoscope will be wedged into an affected lung segment guided by CT scanning. After wedging the bronchoscope, 120ml of sterile 0.09% normal saline will be instilled. All subsequent aliquots will be pooled. Up to 40-60 mL of BAL fluid will be obtained for analysis during each sampling. Alveolar macrophages will be sorted on a fluorescence-activated cell sorter (FACS) Aria III instrument. High-throughput single cell transcriptomic (Drop-seq) data will be processed on Northwestern high-performance computational cluster using Cell Ranger pipeline and post-processed using modified AltAnalyze pipeline.

ELIGIBILITY:
Inclusion Criteria:

* meet 2013 ACR criteria for diagnosis of SSc
* have radiographic evidence for ILD and a forced vital capacity <70% on PFT
* have not taken immune suppression in the last 2 months OR have taken a stable dose of mycophenolate mofetil, rituximab, or prednisone less than or equal to 10 mg for at least 6 months

Exclusion Criteria:

* diagnosis of an overlap syndrome, such as lupus or rheumatoid arthritis
* unable to provide informed consent in English
* currently pregnant or nursing
* current smoker or former smoker (greater than 10 pack years)
* leukopenia
* anemia
* comorbidities of uncontrolled congestive heart failure, cancer not in remission, HIV, or chronic liver disease
* known or suspected infection in the past 3 months
* BMI greater than or equal to 30 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with SSc-ILD will be recruited from the Northwestern University Scleroderma Program.
  Healthy control subjects recruited from the Northwestern community.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2024-03-08 (Actual)

PRIMARY OUTCOMES:
Single-cell RNA-seq analysis | Baseline and 6 months
  Change in alveolar macrophage transcriptome at 6 months, as measured by single cell RNA-sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Cara Gottardi, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States